CLINICAL TRIAL: NCT00533884
Title: Neurocognitive Functioning in Adults With Upper Aerodigestive System Cancers
Brief Title: Neurocognitive Functioning in Patients With Newly Diagnosed Upper Aerodigestive Tract Cancer Receiving Treatment at Henry-Joyce Cancer Clinic
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000565963; P30CA068485 (NIH); VU-VICC-SUPP-0751
Record Dates: First submitted 2007-09-20; First posted 2007-09-24 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Neurocognitive Impairment; Delirium; Esophageal Cancer; Head and Neck Cancer; Lung Cancer
Keywords: delirium; cognitive/functional effects; hypopharyngeal cancer; laryngeal cancer; lip and oral cavity cancer; metastatic squamous neck cancer with occult primary; nasopharyngeal cancer; oropharyngeal cancer; paranasal sinus and nasal cavity cancer; salivary gland cancer; esophageal cancer; non-small cell lung cancer; small cell lung cancer
MeSH Terms: conditions — Delirium; Esophageal Neoplasms; Head and Neck Neoplasms; Lung Neoplasms; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Mouth Neoplasms; Nasopharyngeal Neoplasms; Oropharyngeal Neoplasms; Salivary Gland Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treatment: Patients undergoing treatment for head and neck, lung, and esophagus cancers
  Interventions: Other: Assessment of therapy complications; Other: Neurocognitive assessment; Other: Quality-of-life assessment

INTERVENTIONS:
Other: Assessment of therapy complications — Assessment of neurocognitive function, functional status, symptom prevalence and distress, and mood alterations
Other: Neurocognitive assessment — Assessment of neurocognitive domains: attention/concentration, executive function, verbal learning, verbal memory, verbal fluency
Other: Quality-of-life assessment — Assessment of quality of life using Cantrill's Ladder at baseline and 3 months post-treatment

SUMMARY:
RATIONALE: Gathering information about how often problems with neurocognitive functioning occur in patients with newly diagnosed upper aerodigestive tract cancers may help doctors learn more about the disease.

PURPOSE: This clinical trial is studying neurocognitive functioning in patients with newly diagnosed upper aerodigestive tract cancers receiving treatment at Henry-Joyce Cancer Clinic.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To establish an estimate of the prevalence of baseline neurocognitive impairment prior to initiation of outpatient cancer treatment.
* To establish an estimate of the incidence of neurocognitive impairment during outpatient cancer treatment.
* To describe how neurocognitive functioning changes over time during cancer treatment.

Secondary

* To identify sociodemographic and clinical factors associated with neurocognitive impairment.
* To examine health-related outcomes associated with neurocognitive impairment.

OUTLINE: Patients undergo interview to complete measures of domain-specific neurocognitive functioning, global neurocognitive functioning, subjective neurocognitive functioning, delirium, physical functioning, symptom prevalence and distress, mood states, and medications at baseline before initiation of cancer treatment, at scheduled treatment visits, and at the follow-up visit 3 months after completion of cancer treatment.

Measures of comorbidity, alcohol use, sensory functioning (vision and hearing), and sociodemographic are completed at baseline only. Cancer-related information (diagnosis, staging, and sites of metastasis, if applicable), treatment-related information (planned treatment regimen - chemotherapy and/or radiation therapy), and current medications are obtained at baseline by medical record review.

Health service use and complications are assessed at each scheduled treatment visit and at the 3-month post-treatment follow-up visit. Measures of domain-specific neurocognitive functioning, coping, and quality of life are completed at baseline and at the 3-month follow-up visit.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed solid tumors of the upper aerodigestive system, including cancers of the head and neck, esophagus, or lung
* Receiving treatment at the Henry-Joyce Cancer Clinic at the Vanderbilt-Ingram Cancer Center
* No known brain metastasis

PATIENT CHARACTERISTICS:

* Able to hear, speak, and understand English
* No prior diagnosis of other cancer except basal cell carcinoma

PRIOR CONCURRENT THERAPY:

* No treatment plans including prophylactic cranial irradiation

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed upper aerodigestive system cancers (head and neck, lung, and esophagus)
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2007-10; Primary Completion 2010-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Domain-Specific Neurocognitive Functioning measuring attention, executive functioning, mental processing speed, verbal memory, language, and visuospatial construction at baseline and 3 months after completion of treatment | Baseline and 3 months post-treatment
Global neurocognitive functioning as measured by the Mini-Mental State Examination (MMSE) | Baseline, at each scheduled treatment visit, and at 3 months post-treatment
Self-reported neurocognitive symptoms as measured by the Alertness Behavior Subscale of the Sickness Impact Profile | Baseline, at each scheduled treatment visit, and at 3 months post-treatment
Delirium and delirium symptoms by the NEECHAM Confusion Scale and Confusion Assessment Method (CAM) | Baseline, at each scheduled treatment visit, and at 3 months post-treatment

SECONDARY OUTCOMES:
Alcohol, tobacco, and drug use as measured by the Alcohol Use Disorders Identification Test (AUDIT) | Baseline
Premorbid intellectual functioning as measured by the North American Adult Reading Test (NAART) | Baseline
Functional status measured by the Duke Older Americans Resources and Services (OARS) Activities of Daily Living Scale | Baseline, at each scheduled treatment visit, and at 3 months post-treatment
Symptom prevalence and distress measured using the short form of the Memorial Symptom Assessment Scale (MSASSF) | Baseline, at each scheduled treatment visit, and at 3 months post-treatment
Mood State measured by the Profile of Mood States (POMS-SF) | Baseline, at each scheduled treatment visit, and at 3 months post-treatment
Overall quality of life measured using Cantril's Ladder | Baseline and 3 months post-treatment
Coping measured by the Mini-Mental Adjustment to Cancer Scale (Mini-MAC) | Baseline and 3 months post-treatment
Hospitalizations, emergency department visits, and unscheduled clinic visits | At each scheduled treatment visit and 3 months post-treatment
Falls, injuries, and other complications | At each scheduled treatment visit and 3 months post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Stewart M. Bond, PhD, RN, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (4):
- United States (4):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - MBCCOP - Meharry Medical College - Nashville, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee